CLINICAL TRIAL: NCT07017387
Title: The Effect of Two Different Health Education Methods on Women's HPV Knowledge, Cervical Cancer Health Belief and Screening Programme.
Brief Title: Impact of Education Methods on HPV Knowledge and Screening Behavior
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Principal Investigator, Serpil Özdemir, Associate Professor, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2025-23
Record Dates: First submitted 2025-05-25; First posted 2025-06-12 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Health Education; Motivational Interviewing
Keywords: cervical cancer; motivational interviewing; health education; HPV
MeSH Terms: conditions — Health Education; Uterine Cervical Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 2: Health Education (Experimental): Participants will receive one face-to-face health education session and a brochure, followed by two reminder sessions via phone.
  Interventions: Behavioral: Health education
- Arm 3: Control Group (No Intervention): Participants will receive standard healthcare services. At the end of the study, they will be offered the intervention of their choice.
- Arm 1: Motivational Interviewing-Based Health Education (Experimental): Participants will receive three sessions of face-to-face health education using motivational interviewing techniques through home visits, along with an informational brochure.
  Interventions: Behavioral: Motivational interviewing based health education

INTERVENTIONS:
Behavioral: Motivational interviewing based health education — Participants will receive three sessions of face-to-face health education using motivational interviewing techniques through home visits, along with an informational brochure.
  Arms: Arm 1: Motivational Interviewing-Based Health Education
Behavioral: Health education — Participants will receive one face-to-face health education session and a brochure, followed by two reminder sessions via phone.
  Arms: Arm 2: Health Education

SUMMARY:
The aim of this study is to evaluate the effect of two different health education methods (one based on motivational interviewing) on women's HPV knowledge, cervical cancer health beliefs, and screening behaviors in women aged 30-65. A total of 96 healthy women who are registered at the Incirli Family Health Center in Ankara, meet the inclusion criteria, and volunteer to participate will be randomly assigned to three groups (32 participants per group).

The control group will receive standard healthcare services. The first intervention group will receive three sessions of motivational interviewing-based health education on cervical cancer prevention through home visits, along with an informational brochure. The second intervention group will receive health education and a brochure, followed by a reminder session via phone. At the end of the study, participants in the control group will be offered the intervention of their choice.

DETAILED DESCRIPTION:
This study aims to evaluate the effect of two different health education methods-one based on motivational interviewing-on HPV knowledge, cervical cancer health beliefs, and screening behavior in women aged 30-65. A total of 96 healthy women, registered at the Incirli Family Health Center in Ankara, who meet the inclusion criteria and provide informed consent, will be randomly assigned into three groups of 32 participants each.

The control group will receive standard healthcare services. The first intervention group will receive three face-to-face educational sessions based on motivational interviewing principles on HPV and cervical cancer prevention through home visits, along with an informational brochure. These sessions will occur during Weeks 1, 2, and 3. A final follow-up session to administer FORM II will be held in Week 8.

The second intervention group will receive a single face-to-face educational session on HPV and cervical cancer prevention (Week 1), receive a brochure, and two follow-up reminder sessions via telephone in Weeks 2 and 3. FORM II will be administered in Week 8.

After the study period, participants in the control group will be offered the opportunity to choose and receive one of the two intervention methods. All participants will complete the HPV Knowledge Scale, the Cervical Cancer and Pap Smear Test Health Belief Model Scale, and a VAS for self-assessment.

ELIGIBILITY:
Inclusion Criteria:

* Being between 30 and 65 years of age
* Being literate
* Agreeing to participate in the study
* Being female
* Being married
* Having no history of cervical cancer in first-degree relatives (mother/sister)
* Not having undergone cervical cancer screening in the last five years
* Not having been diagnosed with cancer

Exclusion Criteria:

* Being pregnant or in the postpartum period
* Having been diagnosed with any type of cancer
* Having a hearing or speech impairment, or a mental disorder
* Using medication due to psychotic treatments
* Having undergone a hysterectomy
* Having had cervical cancer screening within the last five years
* Having received all three doses of the HPV vaccine

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-05-09 (Actual); Primary Completion 2025-06-11 (Actual); Study Completion 2025-09-12 (Estimated)

PRIMARY OUTCOMES:
Change in screening behavior | 8 weeks after intervention
  Binary outcome (Yes/No) capturing whether the participant underwent screening during the follow-up period. If Yes, the result is recorded; if No, the reason for non-participation is documented.
Change in Health Belief About Cervical Cancer and Pap Smear as Measured by the Cervical Cancer and Pap Smear Health Belief Model Scale (35 items) | 8 weeks after intervention
  The 35-item scale (Güvenç et al., 2011) has five subscales: Benefits & Motivation (8 items), Barriers (14), Perceived Severity (7), Perceived Susceptibility (3), Health Motivation (3). Responses use a 5-point Likert scale (1 = Strongly disagree to 5 = Strongly agree). Subscale scores are summed; higher scores reflect stronger beliefs, except Barriers, where higher scores indicate more perceived barriers.
Change in HPV Knowledge Score Measured by the 33-item HPV Knowledge Scale | 8 weeks after intervention
  The 33-item HPV Knowledge Scale (Demir & Özdemir, 2019) assesses knowledge of HPV infection, screening, and vaccination. Each item is answered Yes/No/Don't know and scored 1 (for correct) or 0 (for incorrect/unknown). Total scores range 0-33; higher scores indicate greater knowledge.

SECONDARY OUTCOMES:
Change in Self-Rated Knowledge About Cervical Cancer and Screening Assessed by a 0-10 Visual Analog Scale (VAS) | 8 weeks after intervention
  Participants rate their knowledge on a 10-cm VAS anchored at 0 ("No knowledge") and 10 ("Completely knowledgeable").

CONTACTS AND LOCATIONS:
Locations (1):
- Incirli Family Health Center, Ankara, Kecioren, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No